CLINICAL TRIAL: NCT00151086
Title: Phase I/II Evaluation of Oral Estramustine and Oral Vinorelbine on an Intermittent Schedule in Patients With Hormone-Refractory Adenocarcinoma of the Prostate
Brief Title: Oral Estramustine and Oral Vinorelbine in the Treatment of Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2001-050
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Estramustine and Vinorelbine (Experimental): Treatment will consist of 28-day cycles with estramustine at a dose of 140mg orally 3 times per day on days 1-3 and 8-10 and vinorelbine orally on days 2 and 9 beginning at dose 50mg/m^2.
  Interventions: Drug: Estramustine; Drug: Vinorelbine

INTERVENTIONS:
Drug: Estramustine
Drug: Vinorelbine

SUMMARY:
Purpose: This clinical trail will combine the chemotherapy drugs, Estramustine and Vinorelbine (Navelbine), on an intermittent therapy strategy based on PSA response in the treatment of hormone refractory prostate cancer. The investigators will determine the tolerable dose of (oral) vinorelbine in combination with (oral) estramustine, and evaluate the efficacy of this treatment for patients with hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
Hormone Refractory prostate cancer refers to advanced disease in which a patient no longer responds to conventional hormonal treatment. When hormone therapy is no longer successful, chemotherapy is a treatment option. However, current single-agent treatment has shown to have limited benefit. In this clinical trial, investigators are evaluating the effectiveness of combining two chemotherapy drugs, Estramustine and Vinorelbine (Navelbine), in the treatment of hormone refractory prostate cancer. Estramustine has been used in the treatment of prostate cancer for many years. Vinorelbine has shown activity in prostate cancer. In addition, the effect of this treatment on the quality of life of patients will be evaluated as measured using the FACT-P.

ELIGIBILITY:
Inclusion:

* Patients must have a histologic diagnosis of adenocarcinoma of the prostate. (No evidence of brain metastasis or untreated spinal cord compression.)
* Patients on total androgen suppression therapy must undergo nonsteroidal antiandrogen withdrawal and demonstrate at rising PSA (Prostate Specific Antigen) 4 weeks after withdrawal for flutamide and 6 weeks after withdrawal for bicalutamide or nilutamide.
* Patients must have measurable soft tissue disease or evaluable (abnormal bone scan and/or elevated PSA). If PSA is the only evidence of progressive disease it must be greater than or equal to 4ng/mL.
* Adequate bone marrow, renal and liver function
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-2 (a measure of general well being on a scale of 0-5 where 0 represents asymptomatic and 5 represents death)
* Must be at least 18 years of age
* Must have a life expectancy of greater than or equal to 12 weeks

Exclusion:

* Have previously received vinca alkaloid-based cytotoxic chemotherapy or radiation to greater than or equal to 50% of the total bone marrow.
* Evidence of brain metastasis
* Spinal cord compression
* Prior malignancy except for in situ carcinoma, nonmelanoma skin cancer, or adequately treated malignancy that has been inactive for less than 3 years
* Patients with preexisting neuropathy of greater than or equal to grade 2
* Active gastrointestinal disease, or a disorder that alters gastrointestinal motility or absorption

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2001-12; Primary Completion 2004-03 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Tolerable Dose of Vinorelbine in Combination with Estramustine | 180 days post dose
  To determine the tolerable dose of oral vinorelbine in combination with oral estramustine on an intermittent schedule, and describe the toxicities of the regimen. The dose will not be escalated until at least 180 days of cumulative observation of acute toxicity in patients enrolled at a particular dose level.

CONTACTS AND LOCATIONS:
Overall Officials: David C. Smith, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States